CLINICAL TRIAL: NCT05504941
Title: Detection of an Endovascular Treatment Target in Patients With an Acute, Spontaneous Intracerebral Hemorrhage - an EXPLOrative Pilot Study (HemEXPLO)
Brief Title: Detection of an Endovascular Treatment Target in Patients With an Acute, Spontaneous Intracerebral Hemorrhage
Acronym: HemEXPLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-01435; th22Psychogios2
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Intracerebral Hemorrhage; Nontraumatic Intracerebral Hemorrhage
Keywords: Digital Subtraction Angiography (DSA); Hemorrhagic stroke; Hematoma expansion; Cerebral DSA
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke | interventions — Diagnosis

STUDY DESIGN:
Intervention Model Description: Explorative, one-arm, open label trial
Masking Description: A person blinded to all clinical data will assess the primary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Intervention: DSA (Experimental): additional diagnostic cerebral DSA
  Interventions: Diagnostic Test: Diagnostic, cerebral Digital Subtraction Angiography (DSA)

INTERVENTIONS:
Diagnostic Test: Diagnostic, cerebral Digital Subtraction Angiography (DSA) — The DSA is the goldstandard for the visualization of brain vessels. For performing a diagnostic cerebral DSA, the femoral artery of the patient will be punctured in the groin. Over this arterial access a catheter will be advanced under fluoroscopy guidance to the target vessel in the brain. After navigation to the targeted brain vessel, contrast media will be injected over the catheter into the vessel. The efflux of the contrast media will be monitored and visualized with fluoroscopy. The additional radiation to the patient due to the DSA will be approx. 1.1 mSv. The duration of the DSA will be 15 to 20 minutes.

SUMMARY:
This study is to determine if a treatment target for a potential endovascular therapy exists in patients with an acute, spontaneous (non-traumatic) ICH.

DETAILED DESCRIPTION:
Hemorrhagic stroke caused by an intracerebral hemorrhage (ICH) is a common (roughly 15% of all strokes) and devastating disease with high rates of mortality and morbidity. The most important potentially modifiable prognostic factor after acute diagnosis of an ICH is hematoma expansion.

The investigators hypothesize that in hyperacute ICH patients a treatment target can be detected with a diagnostic, cerebral DSA. The DSA is the goldstandard for the visualization of brain vessels. A treatment target would be a vessel from which contrast media extravasates as a sign of an active bleeding. If such a target could be identified, it could lay the rationale for future trials which would evaluate if stopping the bleeding directly at the origin improves patient outcomes. The only intervention in this study is an additional diagnostic cerebral DSA. This study is to determine if a treatment target for a potential endovascular therapy exists in patients with an acute, spontaneous (non-traumatic) ICH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an acute spontaneous ICH based on non-contrast CT
* Time from symptom onset to anticipated start of cerebral DSA of under 3 hours
* Agreement of the treating physician to perform DSA
* Informed consent documented by signature or fulfilling the criteria for emergency consent procedures (deferral of consent)

Exclusion Criteria:

* High probability that the etiology of the bleeding is a ruptured aneurysm, an arteriovenous malformation or an amyloid angiopathy as judged by the treating physician
* Any time critical surgical or minimal invasive intervention is planned
* Evidence of an ongoing pregnancy, a negative pregnancy test is mandatory in all persons of childbearing potential
* Contraindications against the use of iodine contrast media
* Known severe kidney insufficiency (Glomerular filtration rate < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of a treatment target for a potential endovascular therapy (binary endpoint: yes/no) | one time assessment at baseline (duration of the DSA will be 15 to 20 minutes)
  Presence of a treatment target for a potential endovascular therapy (binary endpoint: yes/no). It is defined by a ruptured artery which fulfills the following two criteria:
  1. Extravasate of contrast media into the surrounding tissue, and
  2. Potentially reachable by a (micro-)catheter which can be used for treatment (i.e., local infusion of a procoagulant medication or (temporary) occlusion of the ruptured artery).

CONTACTS AND LOCATIONS:
Overall Officials: Marios-Nikos Psychogios, Prof Dr, Study Director — Department of Neuroradiology, University Hospital Basel; Urs Fischer, Prof Dr, Study Chair — Department of Neurology, University Hospital Basel
Locations (1):
- Department of Neuroradiology, University Hospital Basel, Basel, Switzerland